CLINICAL TRIAL: NCT05544019
Title: A Phase 1, Open-Label, Multicenter, Dose Escalation Study of SGR-1505 as Monotherapy in Subjects With Mature B-Cell Malignancies
Brief Title: Study of SGR-1505 in Mature B-Cell Neoplasms
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Schrödinger, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SGR-1505-101
Record Dates: First submitted 2022-08-19; First posted 2022-09-16 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Mature B-Cell Neoplasm; Non Hodgkin Lymphoma; DLBCL; Waldenstrom Macroglobulinemia; MALT Lymphoma; Follicular Lymphoma; Pediatric-Type Follicular Lymphoma; IRF4 Gene Rearrangement; EBV-Positive DLBCL, Nos; Burkitt Lymphoma; Plasmablastic Lymphoma; High-grade B-cell Lymphoma; Primary Cutaneous Follicle Center Lymphoma; Primary Effusion Lymphoma; Mantle Cell Lymphoma; DLBCL Germinal Center B-Cell Type; Primary Mediastinal Large B Cell Lymphoma; T-Cell/Histiocyte Rich Lymphoma; ALK-Positive Large B-Cell Lymphoma; Primary Cutaneous Diffuse Large B-Cell Lymphoma; Splenic Marginal Zone Lymphoma; Chronic Lymphocytic Leukemia; Nodal Marginal Zone Lymphoma; HHV8-Positive DLBCL, Nos; Lymphoplasmacytic Lymphoma; Duodenal-Type Follicular Lymphoma
Keywords: MALT1; NF-kB; Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Waldenstrom Macroglobulinemia; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Follicular; Pyloric Stenosis, Hypertrophic; Burkitt Lymphoma; Plasmablastic Lymphoma; Lymphoma, Primary Effusion; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation (Experimental): Up to 9 dose levels in total will be evaluated across two dosing schedules. Eligible patients will be assigned to a dose level cohort according to an accelerated titration design that will transition to a traditional 3+3 dose escalation.
  Interventions: Drug: SGR-1505

INTERVENTIONS:
Drug: SGR-1505 — SGR-1505 will be administered orally.

SUMMARY:
The purpose of this study is to evaluate safety and tolerability and to determine the maximum tolerated dose (MTD) or maximum administered dose (MAD) and/or recommended dose (RD) of SGR-1505.

DETAILED DESCRIPTION:
This is a study of SGR-1505, an oral inhibitor of MALT1, in subjects with relapsed/refractory (R/R) B-cell lymphomas to evaluate the safety, pharmacokinetics (PK), pharmacodynamics (PD), maximum tolerated dose (MTD) or maximum administered dose (MAD) and/or recommended dose (RD) of SGR-1505. Exploratory cohorts will evaluate additional PK, PD, preliminary anti-tumor activity, and safety to establish the SGR-1505 RD. A planned amendment will evaluate SGR-1505 in combination with other anti-cancer agents, such as BTK and BCL-2 inhibitors, in patients with specific B-cell malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have a history of histologically or cytologically confirmed mature B-cell malignancy.
* Subject must have measurable or detectable disease according to the applicable disease-specific classification system and meet criteria for initiation of treatment.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Life expectancy ≥ 12 weeks.

Exclusion Criteria:

* The subject is in need of immediate cytoreductive therapy (unless the patient has no remaining treatment choice with potential benefit).
* Subject has previous invasive malignancy in the last 2 years.
* Subject has a known allergy to SGR-1505 or excipients of SGR-1505.
* Subject has symptomatic or active CNS involvement of disease.
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding that would place the participant at increased risk to the use of an investigational drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-04-10 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Nature, severity, and number of incidences of adverse events (AEs), serious AEs (SAEs), and AEs leading to treatment discontinuation. | Throughout the study, up to 2 years.
Nature and number of incidences of dose limiting toxicity (DLT). | The first 21 days.
  A DLT is an AE that requires treatment interruption.

SECONDARY OUTCOMES:
SGR-1505 Maximal Plasma Concentration (Cmax) | Through study completion, up to 2 years.
  Concentrations of SGR-1505 in plasma are measured at various timepoints following its administration to calculate typical exposure/PK parameters, including, but not limited to, the maximal plasma concentration (Cmax).
SGR-1505 Time to Maximal Plasma Concentration (tmax) | Through study completion, up to 2 years.
  Concentrations of SGR-1505 in plasma are measured at various timepoints following its administration to calculate typical exposure/PK parameters, including, but not limited to, the time to maximal plasma concentration (tmax).
SGR-1505 Area Under the Concentration Versus Time Curve (AUC) | Through study completion, up to 2 years.
  Concentrations of SGR-1505 in plasma are measured at various timepoints following its administration to calculate typical exposure/PK parameters, including, but not limited to, the area under the concentration versus time curve (AUC).
Objective Response Rate (ORR) | Throughout the study, up to 2 years.
  Number of patients who have an objective response per response criteria other than stable disease (SD) or progressive disease (PD) to treatment.
Duration of Response (DOR) | Throughout the study, up to 2 years.
  The time from response CR/PR until relapse or death from any cause.
Disease Control Rate | Throughout the study, up to 2 years.
  PR, CR, and SD for 2 post-baseline disease assessments at least 6 weeks apart.

CONTACTS AND LOCATIONS:
Overall Officials: Frank G Basile, M.D., Study Director — Schrodinger Inc.
Locations (36):
- United States (16):
  - Banner Health - MD Anderson Cancer Center, Gilbert, Arizona
  - Christiana Care Hospital - Helen F Graham Cancer Center, Newark, Delaware
  - Napa Research, Pompano Beach, Florida
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Regional Cancer Care Associates, Hackensack, New Jersey
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Weill Cornell, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University, Durham, North Carolina
  - Gabrail Cancer & Research Center, Canton, Ohio
  - The Ohio State University - The James Cancer Hospital, Columbus, Ohio
  - Oregon Health and Science University - Knight Cancer Institute, Portland, Oregon
  - Rhode Island Hospital, Providence, Rhode Island
  - University of Texas Southwestern, Dallas, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- France (2):
  - AP-HP Hôpital Henri-Mondor, Créteil
  - Institut Gustave Roussy, Villejuif
- Italy (5):
  - Azienda Ospedaliera Nazionale SS. Antonio e Biagio e C. Arrigo - Presidio Ospedaliero SS Antonio e Biagio e Cesare Arrigo, Ospedale Civile, Alessandria
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - AOU Citta della Salute e della Scienza di Torino - Ospedale le Molinette, Torino
  - Azienda Ospedaliera - Universitaria Integrata di Verona - Ospedale Borgo Roma, Verona
- Institute of Oncology, ARENSIA Exploratory Medicine, Chisinau, Moldova
- Poland (3):
  - Uniwersyteckie Centrum Kliniczne, Osrodek Badan Klinicznych Wczesnych Faz, Gdansk
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. M. Kopernika w Lodzi, Lodz
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie, Warsaw
- Romania (2):
  - ARENSIA Institutul Oncologic Prof. Dr. Alexandru Trestioreanu Bucuresti, Bucharest
  - ARENSIA Institutul Oncologic Prof. Dr. Ion Chiricuta Cluj Napoca, Cluj-Napoca
- Spain (6):
  - Institut Catala d'Oncologia - L'Hospitalet, Barcelona
  - Hospital Universitario Quironsalud Madrid, Madrid
  - START Madrid - CIOCC, Madrid
  - START Madrid - Hospital Fundacion Jimenez Diaz, Madrid
  - Clinica Universidad de Navarra - Pamplona, Pamplona
  - Hospital Clinico Universitario de Salamanca, Salamanca
- ARENSIA Research Clinic at Harmony Health Clinic, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: No